CLINICAL TRIAL: NCT04861857
Title: Effects of Parmigiano Reggiano on Muscle and Inflammatory Response to 12 Weeks of Eccentric Resistance Training in Older Adults
Brief Title: Effects of Parmigiano Reggiano on Muscle and Inflammatory Response to Eccentric Resistance Training in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PaRMA.2
Record Dates: First submitted 2021-04-23; First posted 2021-04-27 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-01

CONDITIONS: Atrophy, Muscular; Aging; Inflammation; Cholesterol Deposition
MeSH Terms: conditions — Muscular Atrophy; Inflammation | interventions — Whey Proteins

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Parmigiano Reggiano (Experimental): participants will consume 50 g/die of the dietary supplement and undergo to eccentric exercise training 3 times/week
  Interventions: Dietary Supplement: Parmigiano Reggiano
- Whey Protein (Active Comparator): participants will consume 20 g/die of the dietary supplement and undergo to eccentric exercise training 3 times/week
  Interventions: Dietary Supplement: Whey Protein

INTERVENTIONS:
Dietary Supplement: Parmigiano Reggiano — subjects will receive 50 g/die of the dietary supplement
  Arms: Parmigiano Reggiano
Dietary Supplement: Whey Protein — subjects will receive 20 g/die of the dietary supplement
  Arms: Whey Protein

SUMMARY:
Aging is associated with the loss of muscle mass and function (sarcopenia) and reduced tissue regenerative capacity.

Eccentric exercise (ECC) is a model of RET that can be used with the elderly, due to the ability of the muscle to combine high muscle strength production with low energy cost. ECC contractions are significantly more damaging to the muscles and produce greater muscle strength, for these reasons there is a greater risk of inducing muscle damage before the muscle is able to adapt.

Parmigiano Reggiano (PR) has some peculiar bromatological characteristics. The proteins contained in it, and in particular the potentially bioactive peptide sequences, can rapidly provide the amino acids necessary to promote muscle growth and repair during exercise. Furthermore, PR can be an important source of fatty acids, of which a significant amount of short-chain fatty acids (SCFA) which are known to have important clinical effects on body composition and metabolic health and can have a systemic anti-inflammatory effect.

Therefore, the central hypothesize is that PR consumed while being engaged in a RET can provide more energy substrates and improve muscle recovery, redcue inflammatory markers and improve lipid metabolism. To date, no studies have studied its function on recovery from exercise nor in the elderly.

ELIGIBILITY:
Inclusion Criteria:

* age >60 years
* BMI >18 and <30 kg/m2
* stable body weight in the past 3 months
* valid medical certifacate for practice of physical activity

Exclusion Criteria:

* diabetes or pre-diabetes as for ADA guidelines
* chronic diseases (cardiovascular, liver, respiratory, cancer, etc)
* acute inflammatory status
* regular practice of intense physical activity (>2 sessions/week)
* treatment with steroids in the past 3 months
* regular use of >50g/die of Parmigiano Reggiano

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2022-03-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Leg lean Mass | Change from baseline to up to 12 weeks
  kg of lean mass measured via DEXA

SECONDARY OUTCOMES:
inflammatory marker: IL-6 | Change from baseline to up to 12 weeks
  levels of plasma IL-6 (mg/dL)
cholesterol | Change from baseline to up to 12 weeks
  levels of plasma cholesterol (mg/dL)

CONTACTS AND LOCATIONS:
Locations (1):
- Nutrition and Exercise Lab, DSB, University of Padova, Padua, Italy